CLINICAL TRIAL: NCT02760290
Title: Comparison of Extraperitoneal and Intraperitoneal Cesarean Technique: Double Blind Controlled Study
Brief Title: Comparison of Extraperitoneal and Intraperitoneal Cesarean Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Baki Senturk, Pirincipal investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 56
Record Dates: First submitted 2016-03-14; First posted 2016-05-03 (Estimated); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Postpartum Fever; Ileus; Hemorrhage; Pain
Keywords: Forced Expiratory Volume in 1 second; Forced expiratory vital capacity; Peak expiratory flow
MeSH Terms: conditions — Puerperal Infection; Ileus; Hemorrhage; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Extraperitoneal group (Experimental): Extraperitoneal cesarean section will perform after rectus sheat incision and carefully bladder dissecting.
  Interventions: Procedure: Extraperitoneal cesarean section
- Intraperitoneal group (Active Comparator): Conventional transperitoneal cesarean will perform
  Interventions: Procedure: Intraperitoneal cesarean section

INTERVENTIONS:
Procedure: Extraperitoneal cesarean section
  Arms: Extraperitoneal group
Procedure: Intraperitoneal cesarean section
  Arms: Intraperitoneal group

SUMMARY:
Cesarean section will performed via intraperitoneally and extraperitoneally. During postoperative period pain, need for analgesia, respiratory function tests, ileus, bowel movement, discharged time will be compared.

DETAILED DESCRIPTION:
Investigators will compared results intra and extraperitoneal cesarean section. Two groups will determine according to random numbers table. After operations, blood count, C reactive proteins, postoperative temperature, need for analgesia, ileus, bowel movement, mobilization time will compare by blind physician. Abdominal, shoulder and incisional pain at postoperative 0, 6, 12, 18, 24, 30 hours will compared by use visual analog score. Neonatal results and complications also will compare. Investigators and participants will be blind regarding technique.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section for any reasons

Exclusion Criteria:

* Involuntary

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Pain Scores as measured by the Visual Analog Scale | 2 days

SECONDARY OUTCOMES:
Blood count | 2 days
C reactive proteins level | 2 days
Complications | 2 days
Discharge time | 4 days
Forced expiratory volume in 1 second | 2 days
Forced vital capacity | 2 days
Peak expiratory flow | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Baki Şentürk, MD, Study Director — Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Locations (1):
- Zeynep Kamil Maternity and Pediatric Research and Training Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Tappauf C, Schest E, Reif P, Lang U, Tamussino K, Schoell W. Extraperitoneal versus transperitoneal cesarean section: a prospective randomized comparison of surgical morbidity. Am J Obstet Gynecol. 2013 Oct;209(4):338.e1-8. doi: 10.1016/j.ajog.2013.05.057. Epub 2013 May 30. PMID 23727518
- [Result] Chou CY, Liang PC, Chen CA, Lee CN. Cervical abscess with vaginal fistula after extraperitoneal Cesarean section. J Formos Med Assoc. 2007 Dec;106(12):1048-51. doi: 10.1016/S0929-6646(08)60082-0. PMID 18194912
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/23727518
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/18194912